CLINICAL TRIAL: NCT05398705
Title: An Interventional Efficacy and Safety, Phase 2, Double-blind, 3-arm Study to Investigate Orally Administered High/Low-dose Cepharanthine Compared With Placebo in Nonhospitalized Asymptomatic or Mild Adult Participants With COVID-19
Brief Title: Study of Oral High/Low-dose Cepharanthine Compared With Placebo in Non Hospitalized Adults With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: YUNNAN BAIYAO GROUP CO.,LTD (Unknown)
Responsible Party: Principal Investigator, Hai Li, professor of department of gastroenterological division, Renji Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEP-Omicron
Record Dates: First submitted 2022-05-29; First posted 2022-06-01 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Asymptomatic COVID-19
Keywords: Asymptomatic COVID-19; cepharanthine; adult
MeSH Terms: interventions — cepharanthine; Tablets

STUDY DESIGN:
Intervention Model Description: Eligible participants with a confirmed diagnosis of SARS-CoV-2 infection in alternate care site will be randomized (1:1:1) to receive low-dose cepharanthine, high-dose cepharanthine or placebo orally every 8 hours for 5 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose cepharanthine + standardized medical treatment (Experimental): Drug: cepharanthine (tablet) Day 1~5: 20mg, Q8H X 5 days + standardized medical treatment
  Interventions: Drug: Cepharanthine
- High-dose cepharanthine + standardized medical treatment (Experimental): Drug: cepharanthine (tablet) Day 1~5: 40mg, Q8H X 5 days + standardized medical treatment
  Interventions: Drug: Cepharanthine
- placebo+standardized medical treatment (Placebo Comparator): Drug: cepharanthine placebo (tablet) Day 1~5: placebo + standardized medical treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cepharanthine — Low-dose: Day 1~5: 20mg, Q8H X 5 days (60mg/day)+SMT
  Other Names: Low- dose Cepharanthine (tablet)
  Arms: Low-dose cepharanthine + standardized medical treatment
Drug: Placebo — Day 1~5: placebo+SMT
  SMT:standardized medical treatment according to Scheme for Diagnosis and Treatment of 2019 Novel Coronavirus Pneumonia (The 9th Trial Edition) from health commission of China, including bed rest, adequate energy and nutrition, pay attention to water and electrolyte balance to maintain a stable internal environment, closely monitor, antiviral drug and Chinese medicine treatment, etc.
  Other Names: Placebo (tablet)
  Arms: placebo+standardized medical treatment
Drug: Cepharanthine — High-dose: Day 1~5: 40mg, Q8H X 5 days (120mg/day) +SMT
  SMT:standardized medical treatment according to Scheme for Diagnosis and Treatment of 2019 Novel Coronavirus Pneumonia (The 9th Trial Edition) from health commission of China, including bed rest, adequate energy and nutrition, pay attention to water and electrolyte balance to maintain a stable internal environment, closely monitor and Chinese traditional medicine, etc.
  Other Names: High- dose Cepharanthine (tablet)
  Arms: High-dose cepharanthine + standardized medical treatment

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of high/low-dose cepharanthine for the Treatment of COVID-19 in asymptomatic and non-pneumonia mild adult participants with COVID-19 who do not need to be in the hospital, but in alternate care site.

DETAILED DESCRIPTION:
Screening participants will sign the appropriate informed consent form (ICF) prior to completion of any study procedures.

Patients will be randomized to one of three arms, all participants will receive standardized medical treatment (SMT) according to Scheme for Diagnosis and Treatment of 2019 Novel Coronavirus Pneumonia (The 9th Trial Edition) from health commission of China, including bed rest, adequate energy and nutrition, pay attention to water and electrolyte balance to maintain a stable internal environment, closely monitor and Chinese traditional medicine, etc.

* low-dose experimental arm：cepharanthine 60mg/day + SMT
* high-dose experimental arm：cepharanthine 120mg/day + SMT
* placebo control arm：placebo + SMT

The primary outcome measure is the time to viral clearance which defined as first positive nucleic acid test to the date of the first negative test (in two consecutive point). SARS-CoV-2 viral load was detected and quantified by RT-PCR using nasopharyngeal swabs . Ct value>35 for both ORF1ab and N gene was considered as negativity.

ELIGIBILITY:
Inclusion Criteria:

* aged over 16 years old with all genders
* SARS-CoV-2 positive（laboratory-confirmed reverse transcription polymerase chain reaction (RT PCR) test)
* patient or immediate adult family member agrees to participate in this study and signs an informed consent form
* asymptomatic or patients with mild covid-19 symptoms
* confirmed SARS-CoV-2 infection within 5 days prior to randomization

Exclusion Criteria:

* Confirmed SARS-CoV-2 infection within > 5 days prior to randomization
* CT shows pneumonia on admission
* diagnosed as severe or critical COVID-19 before intervention
* has a history of chronic underlying disease and acute exacerbation of that underlying disease at the time of admission
* Females who are pregnant or breastfeeding

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Time to viral clearance | Day 1 through Day 28
  The time to viral clearance was defined as first positive nucleic acid test（or randomization） to the date of the first negative test (in two consecutive point)
SARS-CoV-2 viral load | Day 1 through Day 28
  SARS-CoV-2 viral load was detected and quantified by RT-PCR using nasopharyngeal swabs . Ct value>35 for both ORF1ab and N gene was considered as negativity.

SECONDARY OUTCOMES:
Proportion of participants developing COVID-19 pneumonia | Day 1 through Day 28
Proportion of participants developing severe pneumonia | Day 1 through Day 28
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)of CEP relative to placebo. | Day 1 through Day 28
Number of days from the onset of fever until the temperature drops below 37.3°C | Day 1 through Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Hai Li, MD, Study Director — Department of gastroenterology, Renji Hospital, Shanghai Jiaotong University School of Medicine
Locations (2):
- China (2):
  - Xinhua Hospital Affiliated To Shanghai Jiao Tong University School Of Medicine, Shanghai, Shanghai Municipality
  - Ren Ji Hospital, School of Medicine, Shanghai Jiao TongUniversity, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided
If shared, including protocol, case report form (CRF), Statistical Analysis Plan (SAP), etc.

REFERENCES:
- [Result] Shen Y, Ai J, Lin N, Zhang H, Li Y, Wang H, Wang S, Wang Z, Li T, Sun F, Fan Z, Li L, Lu Y, Meng X, Xiao H, Hu H, Ling Y, Li F, Li H, Xi C, Gu L, Zhang W, Fan X. An open, prospective cohort study of VV116 in Chinese participants infected with SARS-CoV-2 omicron variants. Emerg Microbes Infect. 2022 Dec;11(1):1518-1523. doi: 10.1080/22221751.2022.2078230. PMID 35579892
- [Result] Hammond J, Leister-Tebbe H, Gardner A, Abreu P, Bao W, Wisemandle W, Baniecki M, Hendrick VM, Damle B, Simon-Campos A, Pypstra R, Rusnak JM; EPIC-HR Investigators. Oral Nirmatrelvir for High-Risk, Nonhospitalized Adults with Covid-19. N Engl J Med. 2022 Apr 14;386(15):1397-1408. doi: 10.1056/NEJMoa2118542. Epub 2022 Feb 16. PMID 35172054
- [Derived] Wei J, Liu S, Bian Y, Li L, Qian B, Shen Z, Zhang Y, Abuduaini A, Dong F, Zhang X, Li J, Yu Y, Zhang W, Wang J, Zhai W, Song Q, Zheng Y, Pan W, Yu L, Zhan Q, Zhang N, Zheng J, Pan S, Yao C, Li H. Safety and efficacy of oral administrated cepharanthine in non-hospitalized, asymptomatic or mild COVID-19 patients: a Double-blind, randomized, placebo-controlled trial : Author detials. Sci Rep. 2025 Jan 31;15(1):3875. doi: 10.1038/s41598-024-75891-3. PMID 39890847